CLINICAL TRIAL: NCT00962104
Title: A Double-Blind Placebo-Controlled Asian Study of Atomoxetine Hydrochloride in the Treatment of Adult Patients With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Atomoxetine to Treat Asian Adult Patients With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12107; B4Z-JE-LYEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 40-120 milligrams (mg) taken by mouth, once daily for 10 weeks.
  Other Names: LY139603
  Arms: Atomoxetine
Drug: Placebo — Taken by mouth, once daily for 10 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, the quality of life, and the safety of multiple dosing atomoxetine in Asian adult subjects with attention deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The treatment will be initiated at the lowest dosage 40 milligrams per day (mg/day), and it will be titrated up to 80 mg/day. Patients who are unable to tolerate a dose of at least 80 mg/day through the end of this study will be discontinued. The dosage will be titrated up to a maximum of 120 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for current attention deficit/hyperactivity disorder (ADHD) as well as criteria for a historical diagnosis of ADHD during childhood, both assessed by the Conners' Adult Attention-Deficit/Hyperactivity Disorder Diagnostic Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition at screening
* Patients must have a score of 2 or greater on at least 6 items of either the inattentive or hyperactive/impulsive core subscales at randomization or screening on the rated Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Investigator Rated: Screening Version (CAARS-Inv:SV) 18-item total ADHD symptom score. In addition, their total score on the 18-item total ADHD symptom score must be 20 or greater.
* Patients must have a Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder-Severity score of 4 (moderate symptoms) or greater.
* Patients must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, required by the protocol.
* Patients must possess an educational level and degree of understanding of the language of their country that enables them to communicate suitably with the investigator and study coordinator.
* Patients must be able to swallow capsules.

Exclusion Criteria:

* Patients who meet full DSM-IV-TR diagnostic criteria for any history of bipolar disorder or any history of schizophrenia and other psychotic disorders, or patients who had received injectable sustained-release neuroleptics.
* Patients with depressive disorder who also have a total score of 12 or greater on the Hamilton Depression Rating Scale-17 items at randomization. Patients who have both a current or past history of major depression and received any anti-depression drug therapy within 6 months of screening.
* Patients who meet DSM-IV-TR diagnostic criteria for current anxiety disorder and also patients who require anti-anxiety drug therapy, except for those taking benzodiazepine analogs for anxiety, which need to be limited.
* Patients who have been diagnosed (DSM-IV-TR) with a pervasive developmental disorder.
* Patients who, in the opinion of the investigator, are at serious suicidal risk or serious risk of harming others, or whose score for Item 11 on the Hamilton Depression Rating Scale-17 items is equal or more than 2 at randomization or screening.
* Patients who have received atomoxetine in a prior clinical study.
* Patients with significant medical conditions that are likely to become unstable during the trial or would likely be destabilized by treatment with atomoxetine.
* Patients with a history of allergy to atomoxetine, severe allergies to more than 1 class of medications, or multiple adverse drug reactions.
* Patients who have received treatment within the past 30 days with a drug that has not received regulatory approval for any indication at the time the informed consent document is obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangjin-Gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sungnam-Si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yangsan
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keelung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Background] Westfall PH, Krishen A. Optimally weighted, fixed sequence and gatekeeping multiple testing procedures. J Stat Plan Inference. 2001;99:25-40.
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Riskind JH, Beck AT, Brown G, Steer RA. Taking the measure of anxiety and depression. Validity of the reconstructed Hamilton scales. J Nerv Ment Dis. 1987 Aug;175(8):474-9. doi: 10.1097/00005053-198708000-00005. PMID 3625186
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine: Treatment was started at 40 milligrams (mg) taken by mouth, once daily. The treatment period was 10 weeks, during which the dosage was up-titrated to a maximum of 120 mg by mouth, once daily.
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 195 | 196
Full Analysis Set | 193 (2 participants were excluded because they failed to take the assigned study medication.) | 195 (1 participant was excluded because that participant failed to take the assigned study medication.)
Completed | 155 | 171
Not Completed | 40 | 25
Not completed — Adverse Event | 10 | 3
Not completed — Entry Criteria Not Met | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 10 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 6 | 8
Not completed — Sponsor Decision | 0 | 1
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 193 | 195 | 388
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.1) | 31.7 (7.8) | 32.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 100 | 203
  Male | 90 | 95 | 185
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 193 | 195 | 388
Region of Enrollment [Number; unit: participants]
  Taiwan | 34 | 34 | 68
  Japan | 123 | 124 | 247
  Korea, Republic of | 36 | 37 | 73
Number of Participants with the Cytochrome P450 2D6 (CYP2D6) Genotype [Number; unit: participants] — Genotype characterization was used to determine participants' metabolic status. The number of participants differs from the overall number of baseline participants because either cytochrome P450 2D6 (CYP2D6) was not collected or was not evaluated due to an error.
  participants
    Extensive metabolizer (EM) | 40 | 45 | 85
    Intermediate metabolizer (IM) | 137 | 137 | 274
    Poor metabolizer (PM) | 0 | 0 | 0
    Ultra-rapid metabolizer (UM) | 4 | 2 | 6
Attention-Deficit/Hyperactivity Disorder (ADHD) Subtype Current [Number; unit: participants] — ADHD subtype was classified by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria.
  participants
    Inattentive | 96 | 95 | 191
    Hyperactive/Impulsive | 4 | 4 | 8
    Combined | 93 | 96 | 189
Prior Stimulant Exposure Status [Number; unit: participants]
  Prior Stimulant Exposure - Yes | 43 | 42 | 85
  Prior Stimulant Exposure - No | 150 | 153 | 303
Current Major Depressive Episode Status [Number; unit: participants] — Current (past 2 weeks) major depressive episode status was assessed using the Mini International Neuropsychiatric Interview (MINI), a structured diagnostic interview that assesses psychiatric disorders.
  participants
    Major Depressive Episode - Yes | 4 | 0 | 4
    Major Depressive Episode - No | 189 | 195 | 384
Recurrent Major Depressive Episode Status [Number; unit: participants] — Recurrent major depressive episode status was assessed using the Mini International Neuropsychiatric Interview (MINI), a structured diagnostic interview that assesses psychiatric disorders.
  participants
    Recurrent Major Depressive Episode - Yes | 1 | 0 | 1
    Recurrent Major Depressive Episode - No | 192 | 195 | 387
Current Major Depressive Episode with Melancholic Features Status [Number; unit: participants] — Current (past 2 weeks) major depressive episode with melancholic features status was assessed using the Mini International Neuropsychiatric Interview (MINI), a structured diagnostic interview that assesses psychiatric disorders.
  participants
    Current Major Depressive Episode with - Yes | 2 | 0 | 2
    Current Major Depressive Episode with - No | 191 | 195 | 386
Current Social Phobia (Social Anxiety Disorder [SAD]) Status [Number; unit: participants] — Current (past month) social phobia (SAD) status was assessed using the Mini International Neuropsychiatric Interview (MINI), a structured diagnostic interview that assesses psychiatric disorders.
  participants
    Current Social Phobia (SAD) - Yes | 3 | 4 | 7
    Current Social Phobia (SAD) - No | 190 | 191 | 381
Obsessive-Compulsive Disorder (OCD) Status [Number; unit: participants] — Current (past month) OCD status was assessed using the Mini International Neuropsychiatric Interview (MINI), a structured diagnostic interview that assesses psychiatric disorders.
  participants
    Current OCD - Yes | 1 | 2 | 3
    Current OCD - No | 192 | 193 | 385
Conners' Adult Attention-Deficit Hyperactivity/Disorder Rating Scale-Investigator Rated: Screening V [Mean (Standard Deviation); unit: units on a scale] — Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Investigator Rated: Screening Version (CAARS-Inv:SV) is a scale that assesses symptom severity over past week. Total ADHD symptom score consisted of 18 items (sum of inattention [9 items, range: 0-27] and hyperactivity-impulsivity [9 items, range: 0-27] subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54. Higher scores indicate greater impairment.
  units on a scale | 33.2 (7.7) | 33.9 (7.5) | 33.6 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Investigator Rated: Screening Version (CAARS-Inv:SV) 18-Item Total Attention-Deficit/Hyperactivity Disorder (ADHD) Symptom Score up to 10 Weeks
Description: CAARS-Inv:SV is a scale that assesses symptom severity over past week. Total ADHD symptom score consisted of 18 items (sum of inattention [9 items, range: 0-27] and hyperactivity-impulsivity [9 items, range: 0-27] subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently) for total score range of 0 to 54. Higher scores indicate greater impairment.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline CAARS-Inv:SV result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -14.3 (10.4) | -8.8 (9.6)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline CAARS-Inv:SV 18-Item Total ADHD Symptom score; Least Squares Mean Difference = -5.78, 95% CI 2-sided [-7.66 to -3.91]

2. Secondary Outcome: Change From Baseline in the Adult Attention-Deficit/Hyperactivity Disorder Quality of Life-29 (AAQoL) Scores up to 10 Weeks
Description: Participant-reported outcome measure used to examine disease-specific functional impairments and QoL for adults with ADHD. The domains include work functioning, family relationships, social functioning, activities of daily living (that is, driving, managing finances), and psychological adaptation (that is, life satisfaction and self-esteem). Individual items scored on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). Range of scores for this subscale is 0 to 100. Consistent with the majority of existing QoL measures, higher scores on AAQoL-29 indicate better functioning.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline AAQoL result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 178 | 190
units on a scale | 12.83 (15.91) | 8.20 (14.09)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — First gated secondary outcome measure. A gatekeeper strategy (Westfall and Krishen 2001) controlled experiment-wise type I error for 2 QoL measures. Treatments were compared stepwise until an outcome failed to be significant (p>0.05); Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline AAQoL total score; Slope = 4.76, 95% CI 2-sided [1.97 to 7.56]

3. Secondary Outcome: Change From Baseline in the European Quality of Life Questionnaire-5 Dimensions (EQ-5D) Health State Score up to 10 Weeks
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline EQ-5D result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 178 | 189
units on a scale | 1.4 (20.3) | 1.5 (18.4)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.289, ANCOVA — Second gated secondary outcome measure. A gatekeeper strategy (Westfall and Krishen 2001) controlled experiment-wise type I error for 2 QoL measures. Treatments were compared stepwise until an outcome failed to be significant (p>0.05); Least Squares Mean difference between 2 treatment groups from Type III sum of squares analysis of covariance model:Change=treatment+country+baseline; Least Squares Mean Difference = -1.82, 95% CI 2-sided [-5.20 to 1.56]

4. Secondary Outcome: The Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Investigator Rated: Screening Version (CAARS-Inv:SV) 18-Item Total Attention-Deficit/Hyperactivity Disorder (ADHD) Symptom Score at 10 Weeks
Description: CAARS-Inv:SV assesses symptom severity over past week. Total ADHD symptom score comprises 18 items (sum of inattention [9 items, range: 0-27] and hyperactivity-impulsivity [9 items, range: 0-27] subscales) using a 4-point scale (0=not at all/never to 3=very much/very frequently). Total score range: 0 to 54. Higher scores=greater impairment. Least Squares Mean Value based on mixed model repeated measures analysis with term for baseline, country, visit, treatment, and treatment*visit. Baseline included as a covariate; thus, treatment difference in observed value is same as change from baseline.
Time Frame: 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline CAARS-Inv:SV result were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 190 | 195
units on a scale | 17.24 (0.74) | 23.42 (0.73)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -6.18, 95% CI 2-sided [-8.13 to -4.22]

5. Secondary Outcome: The Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Screening Version (CAARS-S:SV) 18 Item Total Attention-Deficit/Hyperactivity Disorder (ADHD) Symptom Score at 10 Weeks
Description: Participant assessment of symptom severity over past week. Total ADHD symptom score comprises 18 items (sum of inattention [9 items, range: 0-27] and hyperactivity-impulsivity [9 items, range: 0-27] subscales) using 4-point scale (0=not at all/never to 3=very much/very frequently). Total score range: 0 to 54. Higher scores=greater impairment. Least Squares Mean Value based on mixed model repeated measures analysis with term for baseline, country, visit, treatment, and treatment*visit. Baseline included as covariate; thus, treatment difference in observed value is same as change from baseline.
Time Frame: 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline CAARS-S:SV result were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | 16.80 (0.77) | 22.97 (0.75)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -6.18, 95% CI 2-sided [-8.21 to -4.14]

6. Secondary Outcome: Change From Baseline in the Behavior Rating Inventory of Executive Function-Adult Version: Self Report (BRIEF-A:Self Report) Score up to 10 Weeks
Description: A 75-item standardized self-reported measure comprised of 3 subscales. Each item is rated on a 3-point Likert scale (1=behavior never observed to 3=behavior often observed). Behavioral regulation subscale measures one's control over behavior (30-90 total score). Metacognition subscale assesses systematic problem-solving ability while sustaining these task-completion efforts in active working memory (40-120 total score). Global executive composite (GEC) subscale rates participant's GEC in everyday environment (75- 225 total score). Higher subscale ratings=greater perceived impairment.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline BRIEF-A result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 177 | 190
units on a scale
  Raw Behavioral Regulation Index Score | -9.1 (12.4) | -5.5 (10.3)
  Raw Metacognition Index (MI) Score (N=177, 189) | -13.6 (17.3) | -7.5 (13.0)
  Raw Global Executive Composite Score (N=175, 189) | -22.6 (28.8) | -13.0 (22.1)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — This is the p-value for the Raw Behavioral Regulation Index score. Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -3.59, 95% CI 2-sided [-5.73 to -1.45]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — This is the p-value for the Raw MI score. Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -6.29, 95% CI 2-sided [-9.28 to -3.31]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — This is the p-value for the Global Executive Composite Index score. Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -9.76, 95% CI 2-sided [-14.75 to -4.78]

7. Secondary Outcome: Change From Baseline in the Behavior Rating Inventory of Executive Function-Adult Version: Informant (BRIEF-A: Informant) Score up to 10 Weeks
Description: Third-party observer of participant completes 75-item scale. Comprised of 3 subscales. Each item rated on 3-point Likert scale (1=behavior never observed to 3=behavior often observed). Behavioral regulation subscale measures one's control over behavior (30-90 total score). Metacognition subscale assesses systematic problem-solving ability while sustaining these task-completion efforts in active working memory (40-120 total score). Global executive composite (GEC) subscale rates participant's GEC in everyday environment (75-225 total score). Higher subscale ratings=greater perceived impairment.
Time Frame: Baseline, up to 10 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 126 | 133
units on a scale
  Raw Behavioral Regulation Index Score (N=126, 128) | -5.8 (10.7) | -5.0 (10.1)
  Raw Metacognition Index (MI) Score | -7.3 (13.6) | -7.3 (12.8)
  Raw Global Executive Composite Score (N=123, 128) | -13.2 (22.7) | -12.4 (21.6)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.092, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -1.93, 95% CI 2-sided [-4.18 to 0.32]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.272, ANCOVA — This is the p-value for the Raw MI Index score. Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -1.62, 95% CI 2-sided [-4.52 to 1.28]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.153, ANCOVA — This is the p-value for the Raw Global Executive Composite Index score. Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -3.55, 95% CI 2-sided [-8.43 to 1.32]

8. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Attention Deficit/Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) up to 10 Weeks
Description: The CGI-ADHD-S is a single-item clinician rating of the clinician's assessment of the overall severity of the participant's ADHD symptoms in relation to the clinician's total experience with ADHD participants. Measures severity of the participant's overall severity of ADHD symptoms (1=normal, not at all ill to 7=among the most extremely ill participants).
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline CGI-ADHD-S result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | -1.3 (1.2) | -0.8 (1.1)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed using an analysis of covariance (ANCOVA) with term for treatment, country, and baseline value; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-0.67 to -0.27]

9. Secondary Outcome: Clinical Global Impression-Attention Deficit/Hyperactivity Disorder-Improvement Scale (CGI-ADHD-I) up to 10 Weeks
Description: The CGI-ADHD-I is a single-item clinician rating of the clinician's assessment of the participant's improvement in ADHD symptoms in relation to the clinician's total experience with ADHD participants. Measures total improvement (or worsening) of a participant's ADHD symptoms from the beginning of treatment (1=very much improved to 7=very much worsened).
Time Frame: Up to 10 weeks
Population: All randomized participants with an endpoint CGI-ADHD-I value within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 191 | 195
units on a scale | 2.84 (0.98) | 3.28 (0.98)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — Statistical significance was assessed using an analysis of variance (ANOVA) with term for treatment and country

10. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Rating Scale-14 Items (HAMA-14) up to 10 Weeks
Description: Clinician-administered rating scale that assesses severity of anxiety and its improvement (or change) during course of treatment (Hamilton 1959; Riskind et al. 1987). Scale consists of 14 items that provide an overall measure of general anxiety, including psychic anxiety and somatic anxiety. Investigator talked to participant about participant's symptoms over previous week before study visit. Each item is rated on a 5-point scale of 0 (absent) to 4 (very severe). Total score=sum of 14 items and ranges from 0 (normal) to 56 (severe). Higher scores indicate a greater degree of symptom severity.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline HAMA-14 result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 179 | 189
units on a scale | -0.6 (3.8) | -0.7 (3.6)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.869, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Least Squares Mean Difference = -0.05, 95% CI 2-sided [-0.71 to 0.60]

11. Secondary Outcome: Change From Baseline in the Hamilton Depression Rating Scale-17 Items (HAMD-17 Total) up to 10 Weeks
Description: The HAMD-17 was used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present) to 4 (very severe) or a 3-point scale of 0 (not present) to 2 (marked). Higher scores indicate greater symptom severity. The total score is the sum of the scores from HAMD-17 Items 1 through 17. The total score may range from 0 (not at all depressed) to 52 (severely depressed). Higher scores indicate a greater degree of symptom severity.
Time Frame: Baseline, up to 10 weeks
Population: All randomized participants with a baseline and at least 1 post-baseline HAMD-17 result within each treatment group, last observation carried forward (LOCF) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 180 | 189
units on a scale | -0.2 (2.9) | -0.1 (2.8)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.870, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Least Squares Mean Difference = -0.05, 95% CI 2-sided [-0.59 to 0.50]

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/193 | 2/195
Other Adverse Events (participants affected / at risk) | 156/193 | 104/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=193) | Placebo (N=195)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=193) | Placebo (N=195)
Constipation (Gastrointestinal disorders) | 17 (17) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 21 (21) | 5 (6)
Nausea (Gastrointestinal disorders) | 81 (100) | 10 (11)
Vomiting (Gastrointestinal disorders) | 13 (16) | 2 (2)
Fatigue (General disorders) | 10 (10) | 9 (9)
Thirst (General disorders) | 21 (23) | 3 (3)
Nasopharyngitis (Infections and infestations) | 9 (9) | 25 (27)
Weight decreased (Investigations) | 13 (13) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 45 (52) | 2 (2)
Dizziness (Nervous system disorders) | 11 (13) | 3 (3)
Headache (Nervous system disorders) | 24 (25) | 20 (26)
Somnolence (Nervous system disorders) | 29 (32) | 22 (26)
Dysuria (Renal and urinary disorders) | 10 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days